CLINICAL TRIAL: NCT01183611
Title: The Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Health Neonates Born to Mother With Positive for Both HBsAg and HBeAg, Positive for HBsAg But Negative for HBeAg, Negative for HBsAg, HBeAg, HBeAb and HBcAb
Brief Title: The Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Health Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Hong-Xin Pan/ MD, Jiangsu Provincial Center for Diseases Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT008
Record Dates: First submitted 2010-05-10; First posted 2010-08-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Virus Disease; DNA Virus Infections; Hepadnaviridae Infections
Keywords: safety; immunogenicity; HBV vaccine; perinatal transmission
MeSH Terms: conditions — Virus Diseases; DNA Virus Infections; Hepadnaviridae Infections | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A1 (Experimental): health neonates born to mother with positive for both HBsAg and e antigen
  Interventions: Biological: Experimental recombinant hepatitis B vaccine, HBIG
- A2 (Active Comparator): health neonates born to mother with positive for both HBsAg and e antigen
  Interventions: Biological: Active Comparator hepatitis B vaccine
- B1 (Experimental): health neonates born to a mother positive for HBsAg, negative for the hepatitis B e antigen
  Interventions: Biological: Experimental recombinant hepatitis B vaccine, HBIG
- B2 (Active Comparator): health neonates born to a mother positive for HBsAg, negative for the hepatitis B e antigen
  Interventions: Biological: Active Comparator hepatitis B vaccine
- C1 (Experimental): health neonates born to mother with negative for the HBsAg and HBeAg and HBeAb and HBcAb
  Interventions: Biological: Experimental recombinant hepatitis B vaccine
- C2 (Active Comparator): health neonates born to mother with negative for the HBsAg and HBeAg and HBeAb and HBcAb
  Interventions: Biological: Active Comparator recombinant hepatitis B vaccine.
- C3 (Placebo Comparator): health neonates born to mother with negative for the HBsAg and HBeAg and HBeAb and HBcAb
  Interventions: Biological: Placebo Comparator recombinant hepatitis B vaccine

INTERVENTIONS:
Biological: Experimental recombinant hepatitis B vaccine, HBIG — Experimental 10mcg/0.5 ml recombinant hepatitis B vaccine and 200IU HBIG
  Arms: A1; B1
Biological: Active Comparator hepatitis B vaccine — Active Comparator 10mcg/0.5 ml of recombinant hepatitis B vaccine，200IU HBIG
  Arms: A2; B2
Biological: Experimental recombinant hepatitis B vaccine — Experimental 10mcg/0.5 ml of recombinant hepatitis B vaccine
  Arms: C1
Biological: Active Comparator recombinant hepatitis B vaccine. — Active Comparator 10mcg/0.5 ml of recombinant hepatitis B vaccine.
  Arms: C2
Biological: Placebo Comparator recombinant hepatitis B vaccine — Placebo Comparator 10mcg/0.5 ml of recombinant hepatitis B vaccine.
  Arms: C3

SUMMARY:
The primary safety objective of this study is to assess the safety of 10 mcg recombinant hepatitis B vaccine in the Chinese health neonates. The primary immunogenicity objective is to assess the antibody response following 3 doses immunization of the 10 mcg experimental dose and 10 or 5 mcg control dose, Participants will include up to 1740 healthy neonates. This is a randomized, double-blinded, Phase III study. This study is designed to investigate the safety, reactogenicity, and immunogenicity of 10ug recombinant hepatitis B vaccine (yeast). Subjects will be stratified by the mother with positive for both HBsAg and HBeAg, positive for the surface antigen but negative for HBeAg, negative for the HBsAg and HBeAg and HBeAb and HBcAb.

* Stratified 1: There are 180 neonates born to the mother with positive for both HBsAg and HBeAg will be randomized into two groups according to the ratio of 2:1. 120 subjects will receive the 10 mcg experimental vaccine and 60 subjects will receive 10 mcg control vaccine respectively.
* Stratified 2: There are 360 neonates born to the mother with positive for HBsAg but negative for HBeAg will be randomized into two groups according to the ratio of 2:1. 240 subjects will receive the 10 mcg experimental vaccine and 120 subjects will receive 10 mcg control vaccine respectively.
* Stratified 3: There are 1200 neonates born to the mother with negative for the HBsAg and HBeAg and HBeAb and HBcAb will be randomized into 3 groups. 600 of them will receive the 10mcg experimental vaccine. 300 subjects will receive 10mcg control vaccine. And the other 300 subjects will receive 5mcg control vaccine.

The recombinant hepatitis B vaccine will be administered at m0, 1 and 6. Following each immunization, safety will be measured by assessment of adverse events through 30 days following each vaccination, serious adverse events and new-onset chronic medical conditions through 6 months post the final vaccination (Day 180 after last vaccination). For the immunogenicity testing will apply the chemiluminescence immunoassay on serum obtained on the day 0, 210 and 360 after born.

DETAILED DESCRIPTION:
During the early 1980s, human plasma-derived hepatitis B vaccines were developed in China. The production of these vaccines has not been adequate to meet China's need. Since the introduction of recombinant vaccines which can be produced in large quantity, at low cost, the emphasis has been placed on a search for a recombinant hepatitis B vaccine. This vaccine is thought to be safe, immunogenic, particularly in infants born to carrier mothers. Since 1992, the 5mcg recombinant hepatitis B vaccine has been used as one of the vaccines in the expanded immunization programs (People's Republic of China). The 5ug recombinant hepatitis B vaccine (yeast) is efficacious in short time but not to persistent in neonates. The primary safety objective of this study is to assess the safety of 10 mcg recombinant hepatitis B vaccine in the chinese health neonates. The primary immunogenicity objective is to assess the antibody response following 3 doses immunization of the 10 mcg experimental dose and 10, 5 mcg control dose, Participants will include up to 1740 healthy neonates.

The primary safety objective of this study is to assess the safety of 10 mcg recombinant hepatitis B vaccine in the Chinese health neonates. The primary immunogenicity objective is to assess the antibody response following 3 doses immunization of the 10 mcg experimental dose and 10 or 5 mcg control dose, Participants will include up to 1740 healthy neonates. This is a randomized, double-blinded, Phase III study. This study is designed to investigate the safety, reactogenicity, and immunogenicity of 10ug recombinant hepatitis B vaccine (yeast). Subjects will be stratified by the mother with positive for both HBsAg and HBeAg, positive for the surface antigen but negative for HBeAg, negative for the HBsAg and HBeAg and HBeAb and HBcAb.

* Stratified 1: There are 180 neonates born to the mother with positive for both HBsAg and HBeAg will be randomized into two groups according to the ratio of 2:1. 120 subjects will receive the 10 mcg experimental vaccine and 60 subjects will receive 10 mcg control vaccine respectively.
* Stratified 2: There are 360 neonates born to the mother with positive for HBsAg but negative for HBeAg will be randomized into two groups according to the ratio of 2:1. 240 subjects will receive the 10 mcg experimental vaccine and 120 subjects will receive 10 mcg control vaccine respectively.
* Stratified 3: There are 1200 neonates born to the mother with negative for the HBsAg and HBeAg and HBeAb and HBcAb will be randomized into 3 groups. 600 of them will receive the 10mcg experimental vaccine. 300 subjects will receive 10mcg control vaccine. And the other 300 subjects will receive 5mcg control vaccine.

All these neonates will have the vaccination within 24 hours after born. The recombinant hepatitis B vaccine will be administered at m0, 1 and 6. Following each immunization, safety will be measured by assessment of adverse events through 30 days following each vaccination, serious adverse events and new-onset chronic medical conditions through 6 months post the final vaccination (Day 180 after last vaccination). For the immunogenicity testing will apply the chemiluminescence immunoassay on serum obtained on the day 0, 210 and 360 after born.

ELIGIBILITY:
Inclusion Criteria:

1. A group (A1-A2)Subjects born to a mother positive for both HBsAg and hepatitis B e antigen.

   • Healthy male and female full-term (37-42 weeks gestation) neonates (birth to 1 day of age)

   • Subjects with a 5-minute Apgar score ≥ 7.

   • Subjects with temperature <37.1°C on axillary setting

   • Subjects with a birth weight ≥ 2.5 kg.

   • Normal neonatal jaundice.
   * Written informed consent obtained from the parent(s) of the subject.
   * Subjects who the investigator believes that their parent(s) can and will comply with the requirements of the protocol.
2. B group(B1-B2) Subjects born to a mother positive for HBsAg, but negative for the hepatitis B e antigen.

   • Healthy male and female full-term (37-42 weeks gestation) neonates (birth to 1 day of age)

   • Subjects with a 5-minute Apgar score ≥ 7.

   • Subjects with temperature <37.1°C on axillary setting

   • Subjects with a birth weight ≥2.5 kg.

   • Normal neonatal jaundice.

   • Written informed consent obtained from the parent(s) of the subject.

   • Subjects who the investigator believes that their parent(s) can and will comply with the requirements of the protocol
3. C group（C1-C3）Subjects born to a mother negative for HBsAg, hepatitis Be Antigen, antibody to hepatitis B core antigen, antibody to hepatitis B e-antigen.

   * Healthy male and female full-term (37-42 weeks gestation) neonates (birth to 1 day of age)
   * Subjects with a 5-minute Apgar score ≥ 7.
   * Subjects with temperature <37.1°C on axillary setting
   * Subjects with a birth weight ≥ 2.5 kg.
   * Normal neonatal jaundice.
   * Written informed consent obtained from the parent(s) of the subject.
   * Subjects who the investigator believes that their parent(s) can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. A group (A1-A2) Subjects born to a mother positive for both HBsAg and e Antigen.

   Exclusion criteria for the first shot • Subjects born to a mother positive for antibody to HBsAg. • Family history of seizures or progressive neurological disease. • Family history of congenital or hereditary immunodeficiency. • History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.

   • Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

   • Subjects born to a mother had administrated of immunoglobulins and/or any blood products during the pregnancy.

   • Use of any investigational or non-registered product other than the study vaccines since birth, or planned use during the study period.

   • Born to a mother known or suspected to be positive for HIV.
   * Family history of congenital or hereditary immunodeficiency.
   * Children in care.
   * Neonatal jaundice requiring systemic treatment.
   * Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
   * Major congenital defects or serious chronic illness, including perinatal brain damage.
   * Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives Exclusion criteria for the second and third shots
   * Dysgenopathy
   * Any reaction or hypersensitivity to the hepatitis B vaccines.
   * Acute infections
   * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
   * Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

<!-- -->

1. B group (B1-B2) Subjects born to a mother positive for HBsAg, but negative for the hepatitis B e antigen.

   Exclusion criteria for the first shot • Subjects born to a mother positive for antibody to HBsAg or e antigen. • Family history of seizures or progressive neurological disease. • Family history of congenital or hereditary immunodeficiency.

   • History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.

   • Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

   • Subjects born to a mother had administrated of immunoglobulins and/or any blood products during the pregnancy.

   • Use of any investigational or non-registered product other than the study vaccines since birth, or planned use during the study period.

   • Born to a mother known or suspected to be positive for HIV.

   • Family history of congenital or hereditary immunodeficiency.

   • Children in care.

   • Neonatal jaundice requiring systemic treatment.

   • Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

   • Major congenital defects or serious chronic illness, including perinatal brain damage.

   • Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives Exclusion criteria for the second and third shots

   • Dysgenopathy

   • Any reaction or hypersensitivity to the hepatitis B vaccines.

   • Acute infections
   * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.

     3 C group (C1-C3) Subjects born to a mother negative for HBsAg, hepatitis Be Antigen, antibody to hepatitis B core antigen, antibody to hepatitis B e-antigen.

   Exclusion criteria for the first shot

   • Subjects born to a mother positive for antibody to HBsAg, or e antigen, or antibody to B core antigen or antibody to hepatitis B e-antigen.

   • Family history of seizures or progressive neurological disease.

   • Family history of congenital or hereditary immunodeficiency.

   • History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.

   • Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

   • Subjects born to a mother had administrated of immunoglobulins and/or any blood products during the pregnancy.

   • Use of any investigational or non-registered product other than the study vaccines since birth, or planned use during the study period.

   • Born to a mother known or suspected to be positive for HIV.

   • Family history of congenital or hereditary immunodeficiency.

   • Children in care.
   * Neonatal jaundice requiring systemic treatment.
   * Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
   * Major congenital defects or serious chronic illness, including perinatal brain damage.
   * Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives Exclusion criteria for the second and third shots
   * Dysgenopathy
   * Any reaction or hypersensitivity to the hepatitis B vaccines.
   * Acute infections
   * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
   * Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1740 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The immunogenicity of experimental recombinant HBV vaccines in healthy neonates on day 210 | on day 210 after the first dose
  Immunogenicity testing will be chemiluminescence immunoassay on serum obtained on day 210 after first dose
The immunogenicity of experimental recombinant HBV vaccines in healthy neonates on day 360 | on day 360 after the first dose
  Immunogenicity testing will be chemiluminescence immunoassay on serum obtained on day 360 after first dose

SECONDARY OUTCOMES:
To evaluate the safety of recombinant HBV vaccines in the health neonates after first dose | within the first 30 days after first dose
  assessment of adverse events through 30 days following first dose
To evaluate the safety of recombinant HBV vaccines in the health neonates after second dose | within the first 30 days after second dose
  assessment of adverse events through 30 days following second dose
To evaluate the safety of recombinant HBV vaccines in the health neonates after third dose | within the first 30 days after third dose
  assessment of adverse events through 30 days following third dose

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhu FC, Liang ZL, Meng FY, Zeng Y, Mao QY, Chu K, Song XF, Yao X, Li JX, Ji H, Zhang YJ, Li L, Pan HX, Xu K, Dai WM, Zhang WW, Deng F, Wang H, Wang JZ. Retrospective study of the incidence of HFMD and seroepidemiology of antibodies against EV71 and CoxA16 in prenatal women and their infants. PLoS One. 2012;7(5):e37206. doi: 10.1371/journal.pone.0037206. Epub 2012 May 25. PMID 22662137